CLINICAL TRIAL: NCT07189130
Title: The Acute Response of Irisin and Brain-derived Neurotrophic Factor in Blood to Resistance Exercise Load
Brief Title: The Acute Effect of Different Resistance Exercise Loads on Irisin and Brain-derived Neurotrophic Factor in Blood Serum and Plasma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0120-222/2024-2711-3
Record Dates: First submitted 2025-08-19; First posted 2025-09-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: BDNF; Irisin; Resistance Exercise; Stroop Test; Lactate; Healthy Young Adult
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: participants going through exercising or control (Experimental): All participants will do 1 control protocol and 3 resistance exercises protocols. Order of protocols will be randomized.
  Interventions: Other: Exercise: 80% 1 RM with 2 minutes break; Other: Exercise: 80% 1RM with1 minute break; Other: Exercise: accenuated eccentric exercise; Other: Control

INTERVENTIONS:
Other: Exercise: 80% 1 RM with 2 minutes break — Participant will do resistance exercise at 80% 1RM with 2 minutes break, 4 sets of each exercise. Included exercises are lat pull, bench press and leg press.
  Other Names: resistance exercise
Other: Exercise: 80% 1RM with1 minute break — Participant will do resistance exercise at 80% 1RM with 1 minutes break, 4 sets of each exercise. Included exercises are lat pull, bench press and leg press.
  Other Names: resistance exercise
Other: Exercise: accenuated eccentric exercise — Participant will do accenuated eccentric resistance exercise at 80% 1RM in concetric part of movement and 110% 1RM in eccentric part of movement with 2 minutes break, 4 sets of each exercise. Included exercises are lat pull, bench press and leg press.
Other: Control — Timeline of events will be same as in exercise protocol (blood withdrawal and Stroop test), except participants will not do any kind of exercise protocol, instead they will be seating.

SUMMARY:
The aim of this study is to investigate different resistance training loads on BNDF and irisin levels in platelets, blood serum and plasma.

DETAILED DESCRIPTION:
In this study, the investigators will examine how three resistance training protocols acutely affect BDNF levels (in serum, plasma, platelet count, and BDNF per platelet) and irisin levels in blood (plasma). The resistance training protocols will differ in intensity, rest intervals between sets and repetition execution. Blood samples will be collected from participants at four time points: before the start of the protocol, 5 minutes after completion of the final set, 1 hour after completion of the final set, and 3 hours after completion of the final set. In addition, blood lactate levels will be monitored at the same time points. Heart rate will also be recorded (immediately before the start of the protocol and 30 seconds after completion of the final set). A control protocol will also be implemented, in which blood will be collected at the same time points. Data will be collected across five visits to the kinesiology laboratory at the University of Ljubljana, Faculty of Sport. Each visit will last approximately 4 hours, except for the first visit where 1RM will be measured.

ELIGIBILITY:
Inclusion Criteria:

* males between 18 and 30 years
* moderate level of physical activity assessed with IPAQ

Exclusion Criteria:

* injuries
* cardiovascular diseases
* respiratory diseases
* psychiatric diseases
* metabolic diseases
* other neurodegenerative diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males.
Enrollment: 24 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
plasma BDNF | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  BDNF will be determined in blood plasma with ELISA kit.
Irisin | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  Irisin will be measured in blood plasma.
serum BDNF | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  BDNF will be determined in blood serum with ELISA kit.
Platelet count | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  Platelet count in blood will be done.
BDNF per platelet | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  The amount of BDNF per platelet will be calculated.

SECONDARY OUTCOMES:
Lactate | pre, 5 minutes post exercise, 1 hour post exercise, 3 hours post exercise.
  Lactate will be measured in blood.
Stroop test | pre, 15 minutes post exercise.
  Stroop test will be used as an assessment of cognitive functions. The number of read word will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Faculty of Sport, Ljubljana, Slovenia